CLINICAL TRIAL: NCT03939247
Title: Effectiveness of High Frequency Currents (Tecarethérapie) in Patients With Lateral Elbow Tendonopathy
Brief Title: Effectiveness of the "Tecaretherapy" in Patients With Lateral Elbow Tendinopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too difficult to recruit patients
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Christophe Demoulin, Associated Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TECARE
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Tendinopathy
Keywords: elbow; tendinopathy; physiotherapy; exercise; electrotherapy
MeSH Terms: conditions — Tendinopathy; Motor Activity | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients receiving the "Placebo Tecare" will be blinded by using an identical device as in the active group but which cannot provide any current
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Conventional PT treatment (CPT)" (Other): All treatment sessions include massage, eccentric exercises by means of an isokinetic dynamometer and stretching;
  Interventions: Other: CPT
- "CPT + Tecare" (Experimental): All treatment sessions include massage, eccentric exercises by means of an isokinetic dynamometer and stretching (idem CPT group). However, an active Tecaretherapy is also provided during the sessions
  Interventions: Other: Active Tecaretherapy; Other: CPT
- "CPT + Placebo Tecare" (Sham Comparator): All treatment sessions include massage, eccentric exercises by means of an isokinetic dynamometer and stretching (idem CPT group). However, an inactive Tecaretherapy is also provided during the sessions
  Interventions: Other: Inactive Tecaretherapy; Other: CPT

INTERVENTIONS:
Other: Active Tecaretherapy — The "Tecaretherapy": consists of using a specific device providing high frequencies (between 300 kHz and 1 MHz) supposed to accelerate the tissues healing process
  Arms: "CPT + Tecare"
Other: Inactive Tecaretherapy — Inactive "Tecaretherapy": the device will not provide any current.
  Arms: "CPT + Placebo Tecare"
Other: CPT — Conventional physiotherapy treatment (massage, eccentric exercises, stretching)

SUMMARY:
This RCT aims at investigating the effectiveness of the "Tecaretherapy" in patients with lateral elbow tendinopathy.

60 patients will be randomized into one of the following 3 groups:

* "Conventional physiotherapy treatment (CPT)" (massage, eccentric exercises, stretching);
* "CPT + Tecare" (idem CPT group + tecaretherapy during the eccentric exercises)
* "CPT + Placebo Tecare" (idem "CPT + Tecare" group but with an inactive Tecare device) The treatment will include 18 30-minute sessions

DETAILED DESCRIPTION:
This RCT aims at investigating the effectiveness of the "Tecaretherapy" in patients with lateral elbow tendinopathy.

60 patients will be randomized into one of the following 3 groups:

* "Conventional physiotherapy treatment (CPT)" (massage, eccentric exercises by means of an isokinetic dynamometer, stretching);
* "CPT + Tecare" (idem CPT group + Tecaretherapy during the eccentric exercises)
* "CPT + Placebo Tecare" (idem "CPT + Tecare" group but with an inactive "Tecare" device) The treatment will include 18 30-minute sessions.

The "Tecaretherapy" consists in using a specific device providing high frequencies (between 300 kHz and 1 MHz) supposed to accelerate the tissues healing process.

Outcome sessions will be organized at baseline, after the first 9 sessions, at the end of the treatment as well as 3 and 6 months after the initial treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a chronic lateral elbow tendinopathy confirmed by echography

Exclusion Criteria:

Patients:

* with contra-indications for a Tecaretherapy (Pace maker, insuline pump, pregnancy, infection, fever, cancer, thrombophlebitis)
* reporting injections and/or shockwaves in the past (for the tendinopathy)
* with an associated neurogenic dysfunction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
change in the "Patient-Rated Tennis Elbow Evaluation" score | up to 6 months
  This questionnaire, developped for patients with elbow tendinopathy, consists of one part dealing with pain and a second part dealing with function. Each of the 5 items in part 1 is scored using a NRS, ranging from 0 (no pain) to 10 (worst pain imaginable). Part 2 is subdivided into Specific Activities (6 items) and Usual Activities (4 items). The 10 items of part 2 use a scale of 0 (no difficulty) to 10 (unable to perform an activity) to rate function. The total score is the combined score that rates pain and disability of equal importance. The pain score total (out of 50 points) and the functional subscale (60 points for specific activities, plus 40 points for usual activities to give a function subscale out of 100 points /2 to provide the remaining 50%) provide a total score, ranging from 0 (no pain and no functional impairment) to 100 (worst pain imaginable with a very significant functional deficit).

SECONDARY OUTCOMES:
change in pain Intensity | up to 6 months
  0-10 Numeric rating scale (0 = no pain, 10 = worst imaginable pain)
change in pain Pressure thresholds | up to 6 months
  Measured by means of an algometer

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vanderthommen, Prof, Principal Investigator — University of Liege; Bénédicte Forthomme, Prof, Principal Investigator — University of Liege
Locations (1):
- CHU Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No